CLINICAL TRIAL: NCT07103473
Title: Interactive Binocular Treatment (I- BiT) in Adult Patients With Anisometropic Amblyopia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Hamideh Sabbaghi, Assistant Professor, Shahid Beheshti University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IR.SBMU.RETECH.REC.1402.438
Record Dates: First submitted 2024-10-27; First posted 2025-08-05 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-08

CONDITIONS: Amblyopia
MeSH Terms: conditions — Amblyopia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Interactive Binocular Treatment (Active Comparator): Patients in this arm will receive the Interactive Binocular Treatment therapy as an intervention
  Interventions: Device: Interactive Binocular Treatment
- Placebo (Placebo Comparator): Patients in this arm will receive no active treatment
  Interventions: Device: Interactive Binocular Treatment

INTERVENTIONS:
Device: Interactive Binocular Treatment — Patients in the intervention group will be asked to play the games which will be designed based on the Interactive Binocular Treatment System and the patients in the placebo group will be asked to play games without the Interactive Binocular Treatment System.

SUMMARY:
Amblyopia is one of the common, preventable and treatable causes of decreased acuity of one or both eyes without a specific organic cause. Common treatments include optical correction, patching (closing the healthy eye), perceptual learning, and drug treatments. The patient's low cooperation, reduction in effectiveness and long treatment period of common methods have led to the design of new treatments that eliminate these disadvantages, among which binocular vision treatments can be mentioned. The purpose of this study is to apply a new and innovative method under binocular conditions in the treatment of anisometropic amblyopia in adults. In this randomized clinical trial study, 30 people (15 patients in the case group and 15 patients in the control group) aged 18 to 40 years with amblyopia (decrease in best corrected vision worse than 0.3 logarithmic units in one of the eyes or the difference of the corrected minimum visual acuity of two lines between two eyes) in the form of two groups of 15 people (case and control) will be included in the study. Patients will be randomly divided into two groups: case and control. Interactive Binocular Treatment (I-BiT) is used in the case group and usual games without I-BiT system are used as placebo in the other group. For this purpose, the games will be presented in the control group in such a way that the two eyes will not be dissociated and the patient will see all the targets in the same way with his two eyes. I-BiT is a new method for the treatment of amblyopia in which a person plays age-appropriate games using special glasses in a 3D space. The stimuli are shown differently to the two eyes and both eyes are involved in the treatment process. The selection of people in two groups will be such that background variables such as age, sex, as well as the severity of amblyopia or vision loss in the two groups are the same and confounding factors are under control. First, all eye examinations such as measuring visual acuity, lateral vision, checking refractive errors with and without cycloplegic drops, checking the alignment of visual axes, and also checking the anterior and posterior segments of the eye are performed. After the definitive diagnosis of amblyopia, people in both groups will be asked to use the given virtual games in the same way for one month, 5 sessions per week, each session for 30 minutes. In order to control the amount of use of computer games by patients, the duration of time that people use games will be controlled and recorded online using software by design engineers. Patients will be examined before treatment, one month after treatment and also one month after stopping treatment.

ELIGIBILITY:
1. Age range from 18 to 40 years
2. Best corrected visual acuity of 0.3 log units or worse in one eye
3. Cases of mild and moderate anisometropic amblyopia (BCVA≤0.3)

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-12-10 (Estimated); Primary Completion 2025-12-10 (Estimated); Study Completion 2025-12-29 (Estimated)

PRIMARY OUTCOMES:
Best corrected visual acuity | one month
  The changes of the best corrected visual acuity after one month therapy will be measured as the primary outcome measure.

SECONDARY OUTCOMES:
Stereopsis | one month
  The changes of stereopsis will be assessed after one month therapy.

CONTACTS AND LOCATIONS:
Locations (1):
- Hamideh Sabbaghi, Tehran, Tehran Province, Iran

IPD SHARING:
Plan to Share IPD: No